CLINICAL TRIAL: NCT03174119
Title: Luminothérapie Chez Les Patients présentant un état de la Conscience altérée: évaluations Comportementale, de Neuroimagerie et (Neuro)Physiologique.
Brief Title: Light Therapy in Disorders of Consciousness: Behavioral, Neuroimaging and (Neuro)Physiological Assessments.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Olivia Gosseries, Dr, University of Liege
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OGosseries
Record Dates: First submitted 2017-05-16; First posted 2017-06-02 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Disorder of Consciousness
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real light exposition by the mean of Luminette® (Active Comparator): All patients will be exposed to a real light (1500 lux, 470 nm) during the treatment phase, 3 times per day (morning, afternoon and evening) for 60 minutes each via goggles providing light at the eyes level. Meanwhile, different assessments will be performed in order evaluating the potential effects of provided light in comparison to placebo ligh. Patients will be given behavioral assessments (Coma Recovery Scale-Revised, Nociception Coma Scale-Revised, brainstem reflexes,...), physiological (body core temperature, saliva, urine, heart rate, blood sample), neuroimaging and neurophysiological tools (PET, fMRI, TMS-EEG, resting-state and auditory paradigm EEG) before, during and after treatment.
  Interventions: Device: Light therapy - active
- Placebo light exposition by the mean of Luminette® (Placebo Comparator): All patients will also be exposed to a placebo light (80 lux, 470 nm) during the treatment phase, 3 times per day (morning, afternoon and evening) for 60 minutes each via goggles providing light at the eyes level. Meanwhile, different assessments will be performed in order evaluating the potential effects of provided light in comparison to placebo light. Patients will be given behavioral assessments (Coma Recovery Scale-Revised, Nociception Coma Scale-Revised, brainstem reflexes,...), physiological (body core temperature, saliva, urine, heart rate, blood sample), neuroimaging and neurophysiological tools (PET, fMRI, TMS-EEG, resting-state and auditory paradigm EEG) before, during and after treatment.
  Interventions: Device: Placebo light

INTERVENTIONS:
Device: Light therapy - active — Active light will be used for one week, as compared to placebo light.
  Other Names: Real light stimulation
  Arms: Real light exposition by the mean of Luminette®
Device: Placebo light — Placebo light will be used for one week, as compared to real light exposition.
  Arms: Placebo light exposition by the mean of Luminette®

SUMMARY:
In this randomized, double-blind, placebo controlled project, the investigators would like to assess the effect of a specific light, as compared to placebo light, on wakefulness (circadian rhythms, homeostasy, sleep-wake cycle), awareness (perceptual and self consciousness), cognition (attention, memory) and underlying brain activity (electrophysiology and neuroimaging)

DETAILED DESCRIPTION:
The investigators will use behavioral (CRS-R, CAP, actimeter, brainstem reflexes), physiological (body core temperature, saliva, urine, heart rate, blood sample), neuroimaging and neurophysiological tools (PET, fMRI, TMS-EEG, resting-state and auditory paradigm EEG) before, during and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* disorder of consciousness
* 6 weeks post-injury

Exclusion Criteria:

* dysautonomia
* acute illnesses (infections with fever)
* medication that is known to affect circadian rhythmicity (melatonin)
* uncorrected sensorial deficits or documented history of significant neurological, neurosurgical, developpemental or psychiatric disorders
* previously known cerebral lesions prior to the brain's insult that lead to disorder of consciousness
* any contraindication to MRI, EEG, TMS-EEG, or PET (e.g., electronic implanted devices, active epilepsy, external ventricular drain)
* not medically stable

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Changes in the Coma Recovery Scale-Revised scores. | 4 weeks study
  Identify the improvement in sleep-wake cycle and circadian rhythm after the real light therapy exposure, with behavioral analyses and diagnosis through the CRS-R results.

SECONDARY OUTCOMES:
Change in sleep-wake cycles through the Nociception Coma Scale-Revised, after the exposition of real light instead of placebo light. | 4 weeks study
  Identify the improvement in sleep-wake cycle and circadian rhythm after the real light therapy exposure, with behavioral analyses through the NCS-R results.
Change in sleep-wake cycles through the actimetry, after the exposition of real light instead of placebo light. | 4 weeks study
  Identify the improvement in sleep-wake cycle and circadian rhythm after the real light therapy exposure, with behavioral analyses through the arms movements measured with the actimetry.
Change in sleep-wake cycles through the brain metabolism with Positron Emission Tomography, after the exposition of real light instead of placebo light. | 4 weeks study
  Identify the improvement in sleep-wake cycle and circadian rhythm after the real light therapy exposure, with PET scan analyses.
Change in sleep-wake cycles through the hemodynamic function of the brain with functional Magnetic Resonance Imaging, after the exposition of real light instead of placebo light. | 4 weeks study
  Identify the improvement in sleep-wake cycle and circadian rhythm after the real light therapy exposure, with fMRI analyses.
Change in sleep-wake cycles through the electrical activity of the brain with electroencephalography, after the exposition of real light instead of placebo light. | 4 weeks study
  Identify the improvement in sleep-wake cycle and circadian rhythm after the real light therapy exposure, with EEG analyses.
Change in sleep-wake cycles through analyses of melatonine hormone, after the exposition of real light instead of placebo light. | 4 weeks study
  Identify the improvement in sleep-wake cycle and circadian rhythm after the real light therapy exposure, with urine analyses.
Change in sleep-wake cycles through temperature measurements, after the exposition of real light instead of placebo light. | 4 weeks study
  Identify the improvement in sleep-wake cycle and circadian rhythm after the real light therapy exposure, with body core temperature analyses.
Change in the outcomes by the assessment of the Glasgow Outcome Scale Extended, after the study. | 2 years after
  Improvement of the recovery's outcomes after the end of the real light therapy exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Laureys, 1, Study Director — University of Liege

IPD SHARING:
Plan to Share IPD: Undecided